CLINICAL TRIAL: NCT01717573
Title: Randomised Controlled Study to Assess Whether Deferred Stenting in Acute STEMI Patients Might Reduce the Incidence of No-reflow Versus Conventional Treatment with Immediate Stenting
Brief Title: Deferred Stent Trial in STEMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NHS National Waiting Times Centre Board (Other)
Collaborators: British Heart Foundation (Other); University of Glasgow (Other); Health Sciences Scotland (Unknown); Chief Scientist Office, Scottish Government (Unknown)
Responsible Party: Principal Investigator, Colin Berry, Consultant Cardiologist, NHS National Waiting Times Centre Board
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Defer-PG-11-2-28474; NCT01851291 (obsolete NCT alias)
Record Dates: First submitted 2012-10-23; First posted 2012-10-30 (Estimated); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: ST-Elevation Myocardial Infarction
Keywords: STEMI; No-reflow; Primary percutaneous intervention; Deferred stenting
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Deferred stenting (Active Comparator): During primary PCI in STEMI, when TIMI 3 flow has been re-established with guide-wire, aspiration thrombectomy and/or balloon angioplasty, stenting is then deferred for a period of 4-16 hours following reperfusion. During this time, patients remain in the Coronary Care Unit and will receive intravenous tirofiban and subcutaneous low molecular weight heparin (enoxaparin 1 mg/kg)
  Interventions: Procedure: Deferred stenting
- Conventional treatment (Sham Comparator): Conventional treatment in STEMI, with immediate stenting
  Interventions: Procedure: Conventional treatment

INTERVENTIONS:
Procedure: Deferred stenting
  Arms: Deferred stenting
Procedure: Conventional treatment
  Arms: Conventional treatment

SUMMARY:
During primary PCI, stent deployment and post-dilatation are associated with no-reflow. The mechanisms for no reflow include distal embolization of thrombus, enhanced thrombus formation and vascular spasm. No reflow is associated with risk factors such as prolonged duration of ischaemia, heavy thrombus burden, persistent ST elevation and long stent length. ACTIVE HYPOTHESIS: once normal antegrade flow has been re-established with initial aspiration thrombectomy and/or balloon angioplasty at the beginning of primary PCI, compared with usual care with direct stenting, a strategy of deferred stenting for 4 -16 hours to permit the beneficial effects of normalized coronary blood flow and anti-thrombotic therapies will reduce the incidence of no reflow in at-risk STEMI patients. DESIGN: In consecutive STEMI patients with risk factors for no reflow and who have given informed consent, when normal flow has been established (TIMI 3) by initial aspiration thrombectomy and/or balloon angioplasty, participants will be randomized to deferred stenting or usual care with direct stenting. All patients will receive dual anti-platelet therapy. Patients who are randomized to deferred stenting will receive intravenous glycoprotein IIbIIIa inhibitor and anti-coagulation with low molecular weight heparin. Patients who are screened and not eligible to be randomized will be prospectively entered into a registry. Study assessments for feasibility, safety and efficacy will be prospectively performed. An independent clinical event committee will review all serious adverse events. Study endpoints will be subject to core laboratory analyses. The study is intended to inform the design of a larger multicentre clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Rescue PCI
* Prolonged ischaemic time (> 12hours)
* Previous MI
* Age > 65
* Occluded artery (TIMI 0/1) at initial angiography
* Thrombus burden (TIMI grade 2+)
* Long plaque/ stent length (> 24 mm)
* Severe coronary artery disease (e.g calcified artery)
* Small reference vessel diameter (< 2.5 mm)
* Persistent ST-elevation (> 50%) following reperfusion
* Index of microvascular resistance (IMR) > 40

Exclusion Criteria:

* Absence of normal coronary flow (TIMI 3)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2012-11 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Incidence of angiographic no-reflow/ slow-reflow (TIMI flow grade < 3) in the deferred and conventional treatment groups | Asessed during the 1st (both groups) and 2nd procedures (deferred group) (0-16 hours)

SECONDARY OUTCOMES:
Extent of late microvascular obstruction (MVO) assessed by cardiac MRI | MRI 2-5 days post randomisation
Clinical events (hospitalisation for heart failure, re-infarction, cardiac death) | Assessed at index admission and 6-months
Degree of ST-segment resolution on ECG | ECG in cath-lab prior to reperfusion and again 60 mins post-reperfusion
TIMI coronary arter flow grade | At the beginning and end of the first procedure (for both groups) and at the beginning and end of the second procedure in the deferred group
Culprit vessel dimensions (QCA) and thrombus burden | Initial coronary angiogram (and 2nd angiogram in deferred group)
Change in LV ejection fraction | Cardiac MRI 2 days and 6-months post PCI
Index of microvascular resistance (IMR) | Assessed following stent deployment (initial procedure for the conventional group and 2nd procedure for the deferred group)
Corrected TIMI frame count | At the beginning and end of the first procedure (for both groups) and at the beginning and end of the second procedure in the deferred group
Angiographic tissue myocardial blush grade | Angiographic myocardial blush grade at the end of the first procedure (both groups) and at the end of the second procedure in the deferred group
Intra-procedural thrombotic events | Asessed during the 1st (both groups) and 2nd procedures (deferred group) (0-16 hours)
Degree of adverse remodelling (end-systolic and end-diastolic volume index) | Cardiac MRI at 6-months
Final infarct size and myocardial salvage | Assessed from cardiac MRI day 2-5 and cardiac MRI at 6months

OTHER OUTCOMES:
Bleeding | Index hospital admission
  Bleeding events related to vascular access or non-access site bleeding. Bleeding was defined according to the ACUITY criteria: major bleed = intracranial or intraocular bleeding; bleeding at the site of angiography requiring intervention; a hematoma of 5 cm in diameter; a reduction in hemoglobin level of at least 4 g/dL in the absence of overt bleeding or 3 g/dL with a source of bleeding; or transfusion.
Contrast nephropathy | Index hospitalization
  Contrast-induced nephropathy was defined as either a greater than 25% increase of serum creatinine or an absolute increase in serum creatinine of 0•5 mg/dL after a radiographic examination using a contrast agent.

CONTACTS AND LOCATIONS:
Overall Officials: Colin Berry, BSc PhD FRCP FACC, Principal Investigator — Golden Jubilee National Hospital; University of Glasgow
Locations (1):
- Golden Jubilee National Hospital, Clydebank, Glasgow, United Kingdom

REFERENCES:
- [Background] Carrick D, Oldroyd KG, McEntegart M, Haig C, Petrie MC, Eteiba H, Hood S, Owens C, Watkins S, Layland J, Lindsay M, Peat E, Rae A, Behan M, Sood A, Hillis WS, Mordi I, Mahrous A, Ahmed N, Wilson R, Lasalle L, Genereux P, Ford I, Berry C. A randomized trial of deferred stenting versus immediate stenting to prevent no- or slow-reflow in acute ST-segment elevation myocardial infarction (DEFER-STEMI). J Am Coll Cardiol. 2014 May 27;63(20):2088-2098. doi: 10.1016/j.jacc.2014.02.530. Epub 2014 Feb 27. PMID 24583294
- [Derived] Gao H, Aderhold A, Mangion K, Luo X, Husmeier D, Berry C. Changes and classification in myocardial contractile function in the left ventricle following acute myocardial infarction. J R Soc Interface. 2017 Jul;14(132):20170203. doi: 10.1098/rsif.2017.0203. PMID 28747397
- See also: British Heart Foundation — https://www.bhf.org.uk/research
- See also: Institute of Cardiovascular and Medical Sciences, University of Glasgow — http://www.gla.ac.uk/researchinstitutes/icams/